CLINICAL TRIAL: NCT07370597
Title: LUtetium-177 DOsimetry as a Predictive Biomarker of Response in Metastatic Prostate Cancer Patients Treated With PSMA Radioligand THerapy.
Acronym: LUDOPATH
Status: Recruiting | Type: Observational
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IJB-MN-LUDOPATH
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer (Adenocarcinoma)
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- eligible patient will perform SPECT/CT and PSMA PET/CT imaging as per local routin

SUMMARY:
A substantial proportion of patients with mCRPC do not respond to 177Lu-PSMA-RLT. The PSA response to Lu-PSMA was observed in nearly 46% of patients included in VISION trial and 66% in LuPSMA trial (4,5). The response to treatment can be evaluated after two cycles using the PSA or PSMA PET/CT scan. Gafita et al. Data have shown that PSA and PSMA perform equally in assessing response to 177Lu-PSMA treatment, and their changes after two cycles are related to patient survival. After two cycles, patients with no PSA or PSMA response had worse outcomes than those with partial response or stable disease . That means PSA and PSMA changes after two cycles can be used as a surrogate of patient outcome. However, the explanation of disease resistance to 177Lu-PSMA-RLT is not yet fully understood. Inappropriate dose administration might be one of the possible explanations. A dose-response relationship has been established in radiotherapy , making dosimetry a standard of care in conventional radiotherapy. In the radionuclide therapy settings, the dose-response relationship has been reported in a multi-center phase 2 trial on the selective internal radiotherapy in hepatocellular carcinoma. In this context, calculating the absorbed dose to tumour lesions could be an excellent method to individualize radionuclide therapy to achieve a maximal response to treatment. If dosimetry calculations could predict which patients would ultimately respond or not respond to treatment, administered dose and number of 177Lu-PSMA-RLT cycles could be adapted early during the treatment course. In this context, our study aims to analyze if absorbed tumour dose obtained by dosimetry calculations could be used as a biomarker to predict non-response to treatment early after one cycle, as the first step towards treatment dose adaptation of a personalized radionuclide treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Male aged ≥18 years with adenocarcinoma of the prostate.
* Progressive metastatic prostate cancer (progression defined as two consecutive increases of PSA, or progression by bone scan or by RECIST1.1).
* Candidate for 177Lu-PSMA-RLT, with at least one lesion showing significant PSMA uptake (uptake higher than liver physiologic activity).
* Able to start treatment within four weeks of baseline PSMA PET/CT.
* Willing and able to comply with all study requirements

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Progressive metastatic prostate cancer
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Patient-based response defined as a decline of serum PSA ≥50% at 12th weeks (after 2 cycles) after treatment initiation. | 12th week after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided